CLINICAL TRIAL: NCT01557049
Title: Global Postural Reeducation in Chronic Low Back Pain: an Randomized Controlled Trial
Brief Title: Global Postural Reeducation in Chronic Low Back Pain
Acronym: GPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Priscila Maria Mendonca de Almeida Lawand, physical therapeutic, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1324/07
Record Dates: First submitted 2012-03-13; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2010-04

CONDITIONS: Back Pain; Mechanical Low Back Pain
Keywords: chronic low back pain; Postural global reeducation; randomized; physical rehabilitation
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postural Reeducation Group (Experimental): The participants, after obtaining a written informed consent, were randomized for one of the two groups: In the Global Postural Reeducation group (GPR), they were submitted 1 time per week, during 12 weeks, at GPR sessions. The duration of sessions was 60 minutes each, with the same physical Therapist of the study. After the intervention, subjects returned to assessment 3 months after, with the blinded assessor. All the 6 postures from GPR were used during the study. All outcomes measurements, in both groups, were validated for Portuguese language and applicable at baseline, 3 months and 6 months after baseline.
  Interventions: Other: Global Reeducation Group
- Control Group (No Intervention): In the control group, no physical intervention was given during the study. After the study, 6 months after, all participants from control group received the same treatment given in GPR group, according to the Unifesp Ethics Committee orientations. All participants, of both groups, have a doctor from the study, if necessary.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Control Group — No physical intervention was given, patients were treated only with medication if necessary.
  Arms: Control Group
Other: Global Reeducation Group — They were treated with medication if necessary and performed GPR session once a week, during 12 weeks. All the 6 postures from GPR were used during the study.
  Arms: Postural Reeducation Group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a Global Postural Reeducation (GPR) program in subjects with chronic low back pain.

DETAILED DESCRIPTION:
Approximately 80-85% of individuals will experience low back pain during their lifetime. It is one of the major concerns of current health care. There is evidence for the effectiveness of exercise therapy in patients with chronic low back pain. GPR is a physical therapy method developed in France by Philippe Emmanuel Souchard. Although this method is largely used as form of treatment in most countries, few studies showed its clinical effectiveness in chronic low back pain. This is the first randomized controlled trial, with assessor blind that evaluate the GPR effects in chronic low back pain. All outcome measurements are reliability, validated and sensitivity for statistical changes using the Visual Analogic Scale- VAS (0-10cm), Roland Morris Questionary, SF36 (Quality Life Questionary) and Beck Scale (Depression Symptoms).

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years age,
* low back pain (more than 12 weeks) without legs irradiation,
* pain between 3-8 cm on a visual Analogue scale (0-10cm).

Exclusion Criteria:

* fibromyalgia,
* pregnancy,
* osteoporosis severe,
* disc herniation,
* patients who had undergone spinal surgical or physiotherapeutic interventions within 3 months prior to baseline assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain | baseline and two follow-up examinations - after 3 and 6 months from baseline
  The primary outcome of this study was the measurement of pain assessed with 0-10cm Visual Analogue Scale (VAS). They were collected at baseline and two follow-up examinations after 3 and 6 months from baseline.

SECONDARY OUTCOMES:
Change from baseline in function | It was collected at baseline and two follow-up examinations after 3 and 6 months from baseline.
  The secondary outcome included function measured by Roland Morris Questionnaire. It was collected at baseline and two follow-up examinations after 3 and 6 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Priscila Maria Lawand, Author, Principal Investigator — Federal University of São Paulo
Locations (1):
- São Paulo Federal University UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Postural Global Reeducation Society — http://www.sbrpg.com.br/
- See also: São Paulo Federal University — http://www.unifesp.br
- See also: Department of Rheumatology from UNIFESP — http://www.unifesp.br/dmed/reumato